CLINICAL TRIAL: NCT04432324
Title: A Multicenter, Randomized, Open-label Parallel Group Pilot Study to Evaluate Safety and Efficacy of High Dose Intravenous Immune Globulin (IVIG) Plus Standard Medical Treatment (SMT) Versus SMT Alone in Hospitalized Subjects With COVID-19
Brief Title: Study to Evaluate the Safety and Efficacy of High Dose IVIG in Hospitalized Participants With Coronavirus Disease (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC2004; 2020-001696-32 (EudraCT Number)
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: Coronavirus Disease; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous Immune Globulin + Standard Medical Treatment (Experimental): Participants will receive the first intravenous (IV) infusion of IVIG on Day 1 up to a net dose of 2 gram per kilogram (g/kg), based upon participant's (body weight) administered in divided doses as infusions of 500 milligram per kilogram (mg/kg), based upon participant's body weight, over 4 days or 400 mg/kg, based upon participant's body weight, over 5 days. Participants will also receive all standard of care interventions while hospitalized, from Day 1 to Day 29.
  Interventions: Biological: Intravenous Immune Globulin; Drug: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Participants will receive all standard of care interventions required throughout the participant's hospitalization, from Day 1 to Day 29
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Biological: Intravenous Immune Globulin — IVIG Intravenous infusion
  Other Names: Flebogamma DIF
  Arms: Intravenous Immune Globulin + Standard Medical Treatment
Drug: Standard Medical Treatment — SMT

SUMMARY:
The purpose of the study is to determine if high dose Intravenous IVIG plus SMT can reduce the proportion of participants dying or requiring intensive care unit (ICU) admission on or before Day 29 or who are dependent on high flow oxygen devices or invasive mechanical ventilation on Day 29 versus SMT alone in hospitalized participants with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized male or female subject ≥ 18 years of age at time of Screening who is being treated for COVID-19.
2. Has laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by qualitative Polymerase Chain Reaction (PCR) (reverse transcriptase [RT]-PCR), or other commercial or public health assay (of any type) in any specimen during the current hospital admission prior to randomization.
3. COVID-19 illness (symptoms) of any duration with radiographic infiltrates by imaging (Chest X-Ray, Computed tomography (CT) scan, etc.).
4. PaO2/FIO2 ratio > 300 to ≤ 450 mmHg (i.e., arterial oxygen in mmHg divided by fraction inspired oxygen concentration [e.g., 0.21 for room air])
5. Any one of the following related to COVID-19: i. Ferritin > 400 nanogram per milliliter (ng/mL), ii. Lactate dehydrogenase (LDH) > 300 units per liter U/L, iii. D-Dimers > reference range, or iv. C-reactive protein (CRP) > 40 milligram per liter (mg/L).
6. Subject (or a legal representative or a nearest relative or a relative by marriage, as appropriate) provides oral informed consent prior to initiation of any study procedures.

Exclusion criteria:

1. Subject requires invasive mechanical ventilation or ICU admission.
2. Clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator may place the subject at undue medical risk.
3. The subject has had a known (documented) serious anaphylactic reaction to blood, any blood-derived or plasma product or commercial immunoglobulin.
4. Subject has known (documented) hereditary fructose intolerance (HFI).
5. A medical condition in which the infusion of additional fluid is contraindicated.
6. Shock that is unresponsive to fluid challenge and/or multiple vasopressors and accompanied by multiorgan failure considered by the Principal Investigator not able to be reversed.
7. Subject with known (documented) thrombotic complications to polyclonal IVIG therapy in the past.
8. Subject with current or prior (within the past 1 month) myocardial infarction, stroke, deep vein thrombosis, or thromboembolic event.
9. Subject with limitations of therapeutic effort (eg, 'do not resuscitate' status).
10. Female subject who are pregnant or of child-bearing potential with a positive test for pregnancy blood or urine human chorionic gonadotropin (HCG)-based assay at Screening/Baseline.
11. Subject participating in another interventional clinical trial with investigational medical product or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Dying or Requiring ICU Admission | Up to Day 29
Percentage of Participants Who are Dependent on High Flow Oxygen Devices or Invasive Mechanical Ventilation | Day 29

SECONDARY OUTCOMES:
Change from Baseline in National Early Warning Score (NEWS) | Day 1 through Day 29
Time to Clinical Response as Assessed by: NEWS ≤ 2 Maintained for 24 hours | Day 1 through Day 29
Time to Hospital Discharge | Day 1 through Day 29
Duration of ICU Stay | Up to Day 29
Duration of Any Oxygen Use | Day 1 through Day 29
Duration of Mechanical Ventilation | Up to Day 29
Mean Change from Baseline in Ordinal Scale | Day 1 through Day 29
Absolute Value Change from Baseline in Ordinal Scale | Day 1 through Day 29
Length of Time to Clinical Progression | Up to Day 29
Percentage of Participants in Each Severity Category of the 7-point Ordinal Scale | Day 15 and Day 29
Time to Sustained Normalization of Temperature | Day 1 through Day 29
Percentage of Participants with Normalization of Fever | Day 1 through Day 29
Number of Participants who Develop Acute Respiratory Distress Syndrome (ARDS) | Day 29

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Getafe, Getafe
  - Hospital Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No